CLINICAL TRIAL: NCT00005006
Title: Cyclical vs Daily Continuous PTH in Combination With Alendronate vs Alendronate Alone
Brief Title: Parathyroid Hormone (PTH) With Alendronate for Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helen Hayes Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Robert Lindsay, Professor of Clinical Medicine, Helen Hayes Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P50AR039191 (NIH); P50AR039191 (NIH); NIAMS-019; Subproject 5
Record Dates: First submitted 2000-03-24; First posted 2000-03-27 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Osteoporosis
Keywords: Anabolic agent; hPTH; PTH; Parathyroid hormone; Bone mass; Bone turnover; Bone formation; Alendronate; Osteoporosis; Cyclical therapy
MeSH Terms: conditions — Osteoporosis | interventions — Parathyroid Hormone; Alendronate; Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Alendronate alone
  Interventions: Drug: Alendronate
- 2 (Active Comparator): Teriparatide daily plus alendronate
  Interventions: Drug: Alendronate; Drug: Teriparatide
- 3 (Active Comparator): Teriparatide cyclically plus alendronate
  Interventions: Drug: Parathyroid Hormone; Drug: Alendronate; Drug: Teriparatide

INTERVENTIONS:
Drug: Parathyroid Hormone — Alendronate 70mg/week; Teriparatide 20mcg/ day
  Other Names: Fosamax; Forteo
  Arms: 3
Drug: Alendronate — Alendronate 70mg/week
Drug: Teriparatide — Teriparatide 20mcg/day
  Arms: 2; 3

SUMMARY:
This study investigates the effectiveness of parathyroid hormone (PTH) in combination with alendronate, a standard treatment for osteoporosis that blocks or reduces bone loss. We are using alendronate because it may help protect patients against any possible harmful effects of PTH in cortical bone such as the long bones or hip. We are testing two different treatment schedules of PTH-one in which we give PTH daily and one in which we give PTH for 3 out of every 6 months in a cyclical fashion. The entire study is 21 months long; the active treatment period is 18 months with a 6-month followup period.

The main effects we will look for in this study are changes in body chemicals that are signs of bone formation or bone breakdown, and changes in bone density throughout the skeleton. We will randomly assign all study participants, who are women aged 50 and over, to either stay on alendronate alone, receive daily continuous PTH plus alendronate, or receive daily PTH for 3 months out of every 6 for a total of three separate 3-month cycles of PTH plus daily alendronate.

DETAILED DESCRIPTION:
Osteoporosis is a significant disease because it increases the risk of fractures throughout the skeleton, most importantly in the spine and hip regions. The current medications for osteoporosis, which include estrogens, bisphosphonates, raloxifene, and calcitonin, all primarily prevent bone loss, although each may be associated with small bone gains. Another class of drugs, the anabolic drugs, will increase bone formation more substantially, leading to bigger gains in bone mass. One of these, sodium fluoride, clearly increases bone mass but may or may not reduce fracture risk. Another bone-forming agent is human parathyroid hormone (PTH). We and others have demonstrated substantial bone mass gains as well as a reduction in vertebral fracture with the use of PTH administered by daily subcutaneous injection.

The current study seeks to capitalize on the knowledge gleaned about PTH-induced stimulation of bone formation prior to resorption in subjects on antiresorptive therapy such as estrogen or alendronate. In this protocol we have chosen to give PTH by daily subcutaneous injection in the presence of alendronate. We have already shown that with 6 weeks of daily subcutaneous h(1-34)PTH 400 U/day in patients on established alendronate, biochemical indicators of bone formation are substantially increased (30-60 percent), with no stimulation of resorption over this time frame.

We hypothesize that, over 3 months, the combination of PTH plus alendronate will, like the combination of PTH plus hormone replacement therapy, result in increments in bone formation exceeding those of bone resorption. We also theorize that this biochemical profile will be reflected in a greater effect on bone mass than during therapy with alendronate alone, when both formation and resorption are elevated. Furthermore, we believe that the changes over the first 3 months can be repeated over additional discrete 3-months cycles after bone turnover returns to baseline.

Therefore, we plan to study the difference in bone mass and biochemical indicators of bone turnover when, in the presence of established alendronate therapy, we give PTH by daily subcutaneous injection continuously for 15 months (in which bone resorption is elevated substantially for more than half of the time) versus discontinuously in three discrete 3-month cycles (in which bone formation will dramatically exceed bone resorption for the entire treatment period).

The candidates for this study are postmenopausal women who have osteoporosis defined by either bone density and/or prior osteoporotic fracture occurrence and, in addition, have used alendronate for at least 18 months prior to entering into the study. Patients must be over the age of 50.

The entire study is 21 months long; the active treatment period is 18 months with a 6- month followup period. The primary outcomes in this study are biochemistry and bone density throughout the skeleton. We will randomly assign all participants to either remain on alendronate alone, receive daily continuous PTH plus alendronate, or receive daily PTH for 3 months out of every 6, for a total of three separate 3-month cycles of PTH, both with PTH given in addition to daily or weekly alendronate.

ELIGIBILITY:
Inclusion Criteria:

* Approximately 140 postmenopausal women, over 50, who have been on alendronate (at least 35 mg/week) for a period of at least 18 months.
* Lumbar spine or hip T-score at the time of recruitment must be equal to or below -2.5.

Exclusion Criteria:

* All subjects must have primary osteoporosis.
* Subjects cannot be on any other medications known to influence bone metabolism besides alendronate. Subjects can be on Synthroid if TSH is normal.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 1987-09; Primary Completion 2003-02 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lindsay, MD, Principal Investigator — Helen Hayes Hospital; Felicia Cosman, MD, Principal Investigator — Helen Hayes Hospital
Locations (1):
- Helen Hayes Hospital, Clinical Research Center, West Haverstraw, New York, United States